CLINICAL TRIAL: NCT02978508
Title: A Multi-center, Double-blind, Randomized, Parallel-group Study Comparing Permethrin Cream, 5% With Elimite™ in Patients With Active Scabies.
Brief Title: Bio-equivalence Study Comparing Permethrin Cream, 5% With Elimite in Patients With Active Scabies.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAP-8184
Record Dates: First submitted 2016-11-17; First posted 2016-12-01 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — Permethrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Permethrin Cream, 5% (Experimental): Permethrin Cream 5%, topical cream, 60g, maximum of two doses over 28 day treatment duration.
  Interventions: Drug: Permethrin Cream, 5%
- Elimite (Active Comparator): Elimite™ 60g, topical, marketed by Prestium Pharma, Inc. ("Prestium"), the branded subsidiary of Renaissance Pharma, maximum of two doses over 28 day treatment duration.
  Interventions: Drug: Elimite

INTERVENTIONS:
Drug: Permethrin Cream, 5% — Subjects on Test product will receive a maximum of two doses, 60 g each, during the study. The first dose will be applied on Day 1 in an outpatient setting, after the visit to the clinical site (preferably in the evening). The second dose will be applied on Day 14±2 only if retreatment is necessary.
  Arms: Permethrin Cream, 5%
Drug: Elimite — Subjects on RLD will receive a maximum of two doses, 60 g each, during the study. The first dose will be applied on Day 1 in an outpatient setting, after the visit to the clinical site (preferably in the evening). The second dose will be applied on Day 14±2 only if retreatment is necessary.
  Other Names: Permethrin Cream, 5%
  Arms: Elimite

SUMMARY:
This is a multi-center, double-blind, randomized, two arm parallel design study. This study is comprised of two phases: screening and treatment. The screening period will be up to 5 days, followed by the treatment phase of 28±4 days. During the treatment phase subjects will be randomized to receive either test or reference treatments in a double-blind manner in an outpatient setting. Randomization of subjects will be in a 1:1 ratio for the test and reference drug arms and will be stratified by site.

Screening will begin at visit 1, during which eligibility will be determined and prohibited treatments will be discontinued. Randomization will occur following the confirmation of the eligibility criteria at visit 2 (baseline, Day 1) i.e. initiation of treatment phase. The treatment phase will be 28±4 days in duration wherein subject will receive treatment with investigational product (either test or reference) on Day 1 or Baseline (visit 2). Safety and tolerability assessments will be performed on Day 7 (visit 3). Efficacy, safety and tolerability will be assessed on Day 14 (visit 4) followed by the End of study visit on Day 28 (visit 5). If positive identification of scabies is confirmed at Day 14 (visit 4), the subject will be retreated with the second application of the investigational product.

DETAILED DESCRIPTION:
Systemic absorption of permethrin cream is limited to 0.5% during the first 48 hours following dermal application. In these settings, a conventional pharmacokinetic human study to demonstrate that Mayne Permethrin cream (5% w/w) is bioequivalent to the Reference Listed Drug [RLD] Elimite™ is not appropriate.

This is a clinical endpoint bioequivalence (BE) study for a Permethrin Cream, 5% formulation for the treatment of active scabies in comparison to Elimite™ Permethrin cream (5% w/w).

* Test Product: Permethrin Cream, 5%
* Reference Product: Elimite™ marketed by Prestium Pharma, Inc. ("Prestium"), the branded subsidiary of Renaissance Pharma.

The infested person, as well as household members are treated at the same time to prevent re-infestation. In consideration of this recommendation, the household members of the enrolled subject will be examined and treated at the same time as the enrolled subject with an FDA-approved generic Permethrin Cream, 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female subject at least 12 years of age or older.
2. Subject must have a positive identification for mites, eggs, or mite fecal matter by microscopic examination of a skin scraping.
3. Subjects must have at least two of the three following: a) excoriations and inflammatory papules with a typical distribution pattern and localization (webbed spaces of the fingers, flexor surfaces of the wrists, elbows, axillae, belt line, feet, skin surface of external genitalia, or areolae); b) presence of burrows; c) family or contacts with moderate to severe itching which increases during the night.
4. Subjects must be willing to make every effort to immediately disinfect clothes, towels, and linens and all potentially infected household items upon diagnosis of infestation to prevent re-infestation.
5. All household members with prolonged physical contact with the subject must be willing to attend Baseline visit and receive treatment with standard of care if deemed necessary by the Investigator in order to prevent re-infestation of the subject enrolled.
6. Subject or representative must read and sign an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved Informed Consent Form (ICF); for minor subjects (18 years or younger in most states) the parent or legal guardian should sign the ICF and the child will be required to sign the Assent Form that will written in such a way as to be understandable to a child.
7. Subject must be able to apply study product to self. If the subject is a child, then parent/guardian will apply study product to him/her.

Exclusion Criteria:

1. Females who are pregnant as shown in a urine pregnancy test at the Baseline visit, prior to randomization, or lactating, or of childbearing potential (for purpose of this study a female of childbearing potential is considered to be not surgically sterile or postmenopausal for at least 1 year) who are not using or do not agree to use an acceptable form of contraception (oral /implant /injectable /transdermal contraceptives, intrauterine device (IUD), condom, diaphragm, or abstinence) during the study, or who intends to become pregnant during the study; contraceptive method must also be consistent throughout the study.
2. Treatment for scabies <4 weeks prior to enrollment, including permethrin, benzyl alcohol, lindane, crotamiton, malathion, and ivermectin.
3. Use of prohibited medications:

   * Topical or oral scabicidal/antiparasitic treatment including: permethrin, benzyl alcohol, benzyl benzoate, lindane, crotamiton, malathion, ivermectin, precipitated sulfur, albendazole, keratolytic cream, tea tree oil, or oil of the leaves of Lippia multiflora Moldenke within 28 days of visit 2.
   * Systemic corticosteroids (including inhaled steroids) taken within 14 days of visit 2.
   * Topical corticosteroids including hydrocortisone taken within 24 hours of visit 2.
   * Topical antipruritics, including antihistamines within 24 hours of any study visits.
   * Oral antihistamine including diphenhydramine (Benadryl) taken within 24 hours of any study visits.
   * Topical antibiotics including mupirocin taken within 24 hours of any study visits.
4. Patients with immunosuppressive disorders requiring therapy, severe systemic disease, history of HIV infection and/or seizures.
5. Patients with crusted/Norwegian scabies.
6. Presence of underlying skin disease that would obscure evaluation of the papules and burrows associated with scabies infection as determined by the Investigator.
7. Presence of severe cutaneous bacterial or fungal infections requiring therapy (including systemic and topical antibiotics) as determined by the Investigator.
8. Sensitivity or allergy to Permethrin Cream or any of its components, synthetic pyrethroids, pyrethrin, chrysanthemums or ragweed.
9. A recent (less than 1 year) history of alcoholism, drug abuse, or other problems which would likely make the subject unreliable for the study.
10. Participation in another investigational study or using any investigational product within the 30 days prior to the Baseline visit.
11. Participation of family member, or another member of the household (including regular bedmates) in the current study.
12. Total number of bedmates and family members with prolonged physical contact is greater than 6 (including study subject).
13. Any employees of the clinic, investigators, or family members of the study staff.
14. Patients who in the opinion of the Investigator would be non-compliant with the requirements of the study protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phoevos Hughes, JD, Study Director — bioRASI, LLC
Locations (3):
- United States (3):
  - LCC Medical Research Institute, Miami, Florida
  - Southcoast Research Center, Miami, Florida
  - Mid Columbia Research, Richland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Permethrin Cream, 5% | Elimite
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Permethrin Cream, 5% | Elimite | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (15.70) | 36.7 (16.23) | 36.3 (15.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 25 | 66
  Male | 29 | 45 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 51 | 103
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 65 | 66 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Visual Examination of Lesions [Count of Participants; unit: Participants] | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients That Are Identified as Cured.
Description: To demonstrate bioequivalence between Permethrin Cream, 5% (Test) and Elimite™ (Reference) in patients with active scabies.
Time Frame: Day 28
Population: 2 subjects were not included in the per protocol anaylis for the following reasons: 101-036: Subject rinsed off the IP after 6:45 mins of application. As per protocol IP is to be rinsed off after at least 8-14 hours of application.
  103003: Subject's visit 3 and 5 was performed out of allowed visit window period.
Measure: Count of Participants; unit: Participants
Arm/Group | Permethrin Cream, 5% | Elimite
Number analyzed (Participants) | 68 | 70
Participants | 68 | 70

2. Secondary Outcome: Proportion of Patients That Are Identified as Cured.
Description: as for outcome 1
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Permethrin Cream, 5% | Elimite
Number analyzed (Participants) | 68 | 70
Participants | 19 | 21

ADVERSE EVENTS:
Time Frame: 7 months from first subject first visit.
Arm/Group | Permethrin Cream, 5% | Elimite
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 8/70 | 5/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Permethrin Cream, 5% (N=70) | Elimite (N=70)
Nasopharyngitis (Infections and infestations) | 2 | 2
Upper Respiratory tract infection (Infections and infestations) | 0 | 1
Burning Sensation (Nervous system disorders) | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02978508/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02978508/SAP_001.pdf